CLINICAL TRIAL: NCT04487873
Title: COVID-19 Phobia and Quality of Life in Patients With Bronchiectasis During Covid-19 Pandemic
Brief Title: COVID-19 Phobia in Patients With Bronchiectasis During Covid-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Merve Firat, Principal Investigator, Hacettepe University
Other Study IDs: GO 20/602
Record Dates: First submitted 2020-07-23; First posted 2020-07-27 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2020-12

CONDITIONS: Covid19; Bronchiectasis
Keywords: phobia; quality of life; health anxiety
MeSH Terms: conditions — COVID-19; Bronchiectasis; Phobic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bronchiectasis: Having been diagnosed with non-cystic fibrosis bronchiectasis
- Healthy individuals: Healthy individuals without chronic disease

SUMMARY:
In the literature, there are no studies evaluating COVID-19 phobia, quality of life, health anxiety, physical activity level and quality of sleep in patients with bronchiectasis during COVID-19 pandemic. The investigators will evaluate these parameters in patients with bronchiectasis and compare the findings of healthy individuals during COVID-19 pandemic

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with non-cystic fibrosis bronchiectasis
* No acute bronchiectasis exacerbation or infection in the past 2 weeks
* Volunteering to participate in the research

Exclusion Criteria:

* Having a cognitive problem
* Not being literate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients and healthy individuals between 18-60 years old, who are diagnosed with non-cystic fibrosis bronchiectasis, and whose local language is Turkish will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
COVID-19 Phobia | 5 minutes
  COVID-19 phobia was evaluated with COVID-19 Phobia Scale (C19P-S) and total score ranges from 20-100. Lower scores mean better outcome.
Qol | 10 minutes
  Quality of life was evaluated with Nottingham Health Profile

SECONDARY OUTCOMES:
Health anxiety | 10 minutes
  Health anxiety was evaluated with Health Anxiety Inventory
Physical activity | 5 minutes
  Physical activity level was evaluated with International Physical Activity Questionnaire - Short Form (IPAQ-SF)
Quality of sleep | 10 minutes
  Quality of sleep was evaluated with Pittsburgh Sleep Quality Index

CONTACTS AND LOCATIONS:
Overall Officials: Merve Firat, MSc, Principal Investigator — Hacettepe University; Naciye Vardar-Yagli, PhD, Study Director — Hacettepe University; Deniz İnal-İnce, Professor, Study Chair — Hacettepe University; Melda Saglam, PhD, Study Chair — Hacettepe University; Ebru Calik-Kütükcü, PhD, Study Chair — Hacettepe University; Aslıhan Cakmak, MSc, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)